CLINICAL TRIAL: NCT05160168
Title: A Phase 1/2 Study of the Safety, Pharmacokinetics and Anti-Tumor Activity of the Oral KIT Inhibitor THE-630 in Patients With Advanced Gastrointestinal Stromal Tumors (GIST)
Brief Title: A Study of THE-630 in Patients With Advanced Gastrointestinal Stromal Tumors (GIST)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The Sponsor terminated the study due to early dose-limiting toxicities.
Sponsor: Theseus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: THE630-21-101
Record Dates: First submitted 2021-11-22; First posted 2021-12-16 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Gastrointestinal Stromal Tumors (GIST); Neoplasms, Connective Tissue; Neoplasms, Connective and Soft Tissue; Neoplasms by Histologic Type; Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasm; Digestive System Disease; Gastrointestinal Diseases
Keywords: Gastrointestinal Stromal Tumor; GIST; KIT inhibitor; THE-630; THE630; THE 630; GIST TKI; GIST tyrosine kinase inhibitor; GIST treatments; GIST Imatinib relapse; GIST Sunitinib relapse; GIST Regorafenib relapse; GIST Ripretinib relapse; PDGFRA; KIT-mutant GIST; Advanced GIST
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Neoplasms, Connective Tissue; Neoplasms, Connective and Soft Tissue; Neoplasms by Histologic Type; Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Digestive System Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose Escalation (Experimental): Participants with unresectable or metastatic GIST who will receive orally administered THE-630.
  Interventions: Drug: THE-630
- Expansion Cohort 1 (Experimental): Patients with unresectable or metastatic GIST who have progressed on or are intolerant to imatinib, sunitinib, regorafenib and ripretinib who will receive orally administered THE-630 at the recommended Phase 2 dose based on the dose escalation phase.
  Interventions: Drug: THE-630
- Expansion Cohort 2 (Experimental): Patients with unresectable or metastatic GIST who have progressed on or are intolerant to imatinib, sunitinib and 0-1 additional lines of therapy in the advanced/metastatic setting, who will receive orally administered THE-630 at the recommended Phase 2 dose based on the dose escalation phase.
  Interventions: Drug: THE-630
- Expansion Cohort 3 (Experimental): Patients with unresectable or metastatic GIST who have progressed on or are intolerant to imatinib (including in the adjuvant setting) and who have not received additional systemic therapy for advanced GIST, who will receive orally administered THE-630 at the recommended Phase 2 dose based on the dose escalation phase.
  Interventions: Drug: THE-630

INTERVENTIONS:
Drug: THE-630 — Oral THE-630 administered once daily in a continuous regimen

SUMMARY:
This study will assess the safety, efficacy, and pharmacokinetics of THE-630 in participants with advanced gastrointestinal stromal tumors (GIST).

DETAILED DESCRIPTION:
The drug being tested in this study is called THE-630, an orally administered KIT tyrosine kinase inhibitor. The study will be conducted in two parts: a dose escalation phase, followed by an expansion phase. The patient population of the initial dose escalation phase (Phase 1) of the trial will include patients with unresectable or metastatic GIST. Patients must have disease progression on or be intolerant to imatinib therapy and have also received at least 1 of the following: sunitinib, regorafenib, ripretinib, or avapritinib. The primary objective of the dose escalation phase is to determine the safety profile of oral THE-630, including the dose limiting toxicities (DLTs), maximum tolerated dose (MTD), and the recommended Phase 2 dose (RP2D).

Once a recommended dose has been determined in the escalation phase, the expansion phase (Phase 2) will enroll 3 cohorts of patients with unresectable or metastatic GIST defined by prior therapy:

* Cohort 1: Patients with unresectable or metastatic GIST who have progressed on or are intolerant to imatinib, sunitinib, regorafenib and ripretinib (≥5th Line).
* Cohort 2: Patients with unresectable or metastatic GIST who have progressed on or are intolerant to imatinib, sunitinib and 0-1 additional lines of therapy in the advanced/metastatic setting (3rd-4th Line).
* Cohort 3: Patients with unresectable or metastatic GIST who have progressed on or are intolerant to imatinib (including in the adjuvant setting) and who have not received additional systemic therapy for advanced GIST (2nd Line).

The safety and tolerability of orally administered THE-630 will continue to be assessed in the expansion cohorts. However, the primary objective of the expansion component of the trial is to evaluate the anti-tumor activity of THE-630 in these GIST patient populations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient ≥18 years of age.
2. For Dose Escalation Phase Cohorts (Phase 1):

   1. Have histologically- or cytologically-confirmed unresectable or metastatic GIST.
   2. Have progressed on or are intolerant to imatinib therapy and have also received at least 1 of the following: sunitinib, regorafenib, ripretinib, or avapritinib.
3. For Expansion Phase Cohorts (Phase 2):

   1. Cohort 1:

      * Have histologically- or cytologically confirmed unresectable or metastatic GIST.
      * Have progressed on or are intolerant to imatinib, sunitinib, regorafenib and ripretinib.
   2. Cohort 2:

      * Have histologically- or cytologically confirmed unresectable or metastatic GIST.
      * Have progressed on or are intolerant to imatinib and sunitinib. Patients in this cohort are allowed to have received up to 1 additional line of therapy in the advanced/metastatic setting.
   3. Cohort 3:

      * Have histologically- or cytologically confirmed unresectable or metastatic GIST.
      * Have progressed on or are intolerant to imatinib (including in the adjuvant setting).
      * Have not received additional systemic therapy for advanced GIST.
4. Have at least 1 measurable lesion as defined by modified RECIST 1.1.
5. Have archival or new tumor biopsy tissue available to submit for mutational testing. Patients without appropriate archival tissue available may be discussed with the study Medical Monitor and approved for enrollment on a case-by-case basis.
6. Have Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2.
7. Adequate renal and hepatic function as defined by the protocol.
8. Adequate bone marrow function as defined by the protocol.
9. For female patients of childbearing potential, have a negative serum or urine beta human chorionic gonadotropin (β-hCG) pregnancy test within 7 days prior to the first dose of study drug.

   o Note: female patients of nonchildbearing potential (postmenopausal; hysterectomy; bilateral salpingectomy; or bilateral oophorectomy) do not require a pregnancy test.
10. Female patients of childbearing potential must agree to abstain from heterosexual intercourse or use a highly effective form of contraception with their sexual partners as defined in the study protocol. Male patients with partners of childbearing potential must agree that they will abstain from heterosexual intercourse or use condoms and their partners will use highly effective contraceptive methods as defined in the study protocol.
11. All toxicities from prior therapy have resolved to Grade ≤1 according to NCI CTCAE v5.0, or have resolved to baseline, at the time of first dose of study drug. Note: treatment-related Grade >1 alopecia, treatment related Grade 2 peripheral neuropathy, and treatment-related Grade 2 hypothyroidism on a stable dose of thyroid hormone replacement therapy are allowed if deemed irreversible.
12. Patient or legal guardian, if permitted by local regulatory authorities, signed and dated informed consent indicating that the patient has been informed of all pertinent aspects of the study.
13. Willingness and ability to comply with scheduled visits and study procedures.

Exclusion Criteria:

1. Received systemic anticancer therapy (including cytotoxic chemotherapy, investigational agent, antineoplastic monoclonal antibodies, or immunotherapy) less than 5 half-lives or 14 days (whichever is shorter) prior to the first dose of study drug.
2. Patients known to be both KIT and PDGFRA wild-type.
3. Received radiotherapy within 14 days prior to the first dose of study drug.
4. Major surgical procedure within 28 days of the first dose of study drug. Minor surgical procedures such as central venous catheter placement or minimally invasive biopsy are allowed.
5. Have known untreated or active central nervous system metastases.
6. 12-lead electrocardiogram (ECG) demonstrating QT interval corrected by Fridericia's formula (QTcF) >470 msec at screening, or history of long QTc syndrome.
7. Have significant, uncontrolled, or active cardiovascular disease, including, but not restricted to:

   * Myocardial infarction (MI) within 6 months prior to the first dose of study drug
   * Unstable angina within 6 months prior to first dose of study drug
   * Symptomatic congestive heart failure (New York Heart Association classes II-IV) within 6 months prior to first dose of study drug
   * Clinically significant, uncontrolled atrial arrhythmia (as determined by the Investigator)
   * Any history of ventricular arrhythmia
   * Cerebrovascular accident or transient ischemic attack within 6 months prior to first dose of study drug
   * Uncontrolled hypertension at study entry. Patients with hypertension should be under treatment on study entry to control blood pressure.
8. Have an active uncontrolled infection, including, but not limited to, the requirement for intravenous antibiotics.
9. Patients with a known allergy or hypersensitivity to any component of the study drug. Patients with a history of Stevens-Johnson syndrome on a prior tyrosine kinase inhibitor (TKI) are excluded.
10. Any active bleeding excluding hemorrhoidal or gum bleeding.
11. For patients with a known human immunodeficiency virus (HIV) infection, have CD4+ T-cell counts <350 cells/uL or history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection within the past 12 months. Patients with HIV infection should be on established antiretroviral therapy (ART) for at least 4 weeks and have an HIV viral load less than 400 copies/mL prior to enrollment.
12. Has known active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, as evidenced by detectable viral load (HBV-DNA or HCV-RNA, respectively). Risk of HBV reactivation should be considered in all patients and the need for anti-HBV prophylaxis should be carefully assessed. Patients with chronic HBV infection with history of active disease who meet the criteria for anti HBV therapy should be on a suppressive antiviral therapy to be eligible for enrollment. Patients who are HCV Ab positive but HCV RNA negative due to prior treatment or natural resolution are eligible. Patients on concurrent HCV treatment at the time of enrollment are allowed if HCV RNA negative.
13. Pregnant or breastfeeding.
14. Malabsorption syndrome or other illness that could affect oral absorption.
15. Patients with prior or concurrent malignancies other than GIST are allowed, except in the case where, in the opinion of the Investigator, the natural history or treatment of the other malignancy has the potential to interfere with the safety or efficacy assessment of the study drug.
16. Have any condition or illness that, in the opinion of the Investigator, might compromise patient safety or interfere with the evaluation of the safety of the drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stew Kroll, Study Director — Theseus Pharmaceuticals (a subsidiary of Concentra Biosciences)
Locations (7):
- United States (7):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Oregon Health & Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Escalation (3 mg Once Daily): Patients with unresectable or metastatic GIST who received orally administered THE-630 (3 mg) once daily in a continuous regimen (28-day cycles).
- Dose Escalation (4 mg Once Daily): Patients with unresectable or metastatic GIST who received orally administered THE-630 (4 mg) once daily in a continuous regimen (28-day cycles).
- Dose Escalation (6 mg Once Daily): Patients with unresectable or metastatic GIST who received orally administered THE-630 (6 mg) once daily in a continuous regimen (28-day cycles).
- Dose Escalation (9 mg Once Daily): Patients with unresectable or metastatic GIST who received orally administered THE-630 (9 mg) once daily in a continuous regimen (28-day cycles).
- Dose Escalation (12 mg Once Daily): Patients with unresectable or metastatic GIST who received orally administered THE-630 (12 mg) once daily in a continuous regimen (28-day cycles).
- Dose Escalation (18 mg Once Daily): Patients with unresectable or metastatic GIST who received orally administered THE-630 (18 mg) once daily in a continuous regimen (28-day cycles).
- Dose Escalation (27 mg Once Daily): Patients with unresectable or metastatic GIST who received orally administered THE-630 (27 mg) once daily in a continuous regimen (28-day cycles).
- Expansion Cohort 1: Patients with unresectable or metastatic GIST who have progressed on or are intolerant to imatinib, sunitinib, regorafenib and ripretinib who will receive orally administered THE-630 (once daily in a continuous regimen) at the recommended Phase 2 dose based on the dose escalation phase.
- Expansion Cohort 2: Patients with unresectable or metastatic GIST who have progressed on or are intolerant to imatinib, sunitinib and 0-1 additional lines of therapy in the advanced/metastatic setting, who will receive orally administered THE-630 (once daily in a continuous regimen) at the recommended Phase 2 dose based on the dose escalation phase.
- Expansion Cohort 3: Patients with unresectable or metastatic GIST who have progressed on or are intolerant to imatinib (including in the adjuvant setting) and who have not received additional systemic therapy for advanced GIST, who will receive orally administered THE-630 (once daily in a continuous regimen) at the recommended Phase 2 dose based on the dose escalation phase.
Period: Overall Study
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily) | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Started | 3 | 7 | 3 | 3 | 3 | 7 | 6 | 0 | 0 | 0
Completed | 3 | 7 | 3 | 3 | 3 | 7 | 6 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in the Expansion cohorts, as the study was terminated by the Sponsor due to dose-limiting toxicities prior to initiation of the Expansion phase (Phase 2) of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily) | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3 | Total
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 7 | 6 | 0 | 0 | 0 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
  Between 18 and 65 years | 2 | 6 | 2 | 3 | 1 | 4 | 2 |  |  |  | 20
  >=65 years | 1 | 1 | 1 | 0 | 2 | 3 | 4 |  |  |  | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (13.01) | 57.7 (10.66) | 57.7 (15.04) | 49.0 (6.00) | 62.7 (9.29) | 64.6 (9.07) | 60.8 (18.32) |  |  |  | 59.3 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 1 | 3 | 4 |  |  |  | 15
  Male | 2 | 5 | 1 | 1 | 2 | 4 | 2 |  |  |  | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 0 | 0 | 1 |  |  |  | 2
  Not Hispanic or Latino | 3 | 7 | 2 | 3 | 3 | 7 | 5 |  |  |  | 30
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 1 | 0 |  |  |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 0 | 0 | 0 |  |  |  | 1
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 0 |  |  |  | 1
  White | 3 | 6 | 3 | 3 | 2 | 6 | 6 |  |  |  | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 7 | 3 | 3 | 3 | 7 | 6 |  |  |  | 32

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation (Phase 1): Safety Analysis - Number of Participants With Treatment-emergent Adverse Events (TEAEs) as Assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Time Frame: Up to 24 months after first dose
Population: Full Analysis Set, which includes all patients who were enrolled and received at least 1 dose of THE-630.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 7 | 6
Participants | 3 | 7 | 3 | 3 | 3 | 7 | 6

2. Primary Outcome: Dose Escalation (Phase 1): Safety Analysis - Number of Participants With Dose-limiting Toxicities (DLTs) Following Oral Administration of THE-630
Time Frame: 28 days
Population: DLT-Evaluable Analysis Set (Phase 1 only), which includes patients enrolled in the Dose Escalation (Phase 1) portion who completed at least 75% of the planned total dose during Cycle 1 (DLT evaluation period, i.e. 21 of 28 days) and patients who experienced a protocol-defined DLT, regardless of dosing adherence in Cycle 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 3 | 3 | 6
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 2

3. Primary Outcome: Dose Escalation (Phase 1): Safety Analysis - Maximum Tolerated Dose (MTD) of Orally Administered THE-630
Description: The MTD is defined as the highest dose at which ≤1 of 6 DLT-assessment eligible patients experience a DLT within the first 28 days of treatment (end of Cycle 1).
Time Frame: 28 days
Population: as for outcome 2
Measure: Number; unit: mg
Groups:
- Dose Escalation (3 mg to 27 mg Once Daily): Patients with unresectable or metastatic GIST who received orally administered THE-630 (3 mg, 4 mg, 6 mg, 9 mg, 12 mg, 18 mg, or 27 mg) once daily in a continuous regimen (28-day cycles).
Arm/Group | Dose Escalation (3 mg to 27 mg Once Daily)
Number analyzed (Participants) | 27
mg | NA — The MTD could not be identified because (1) the 18 mg once daily dose level did not enroll 6 DLT-assessment eligible patients and (2) the 27 mg once daily dose level was shown to exceed the MTD.

4. Primary Outcome: Dose Escalation (Phase 1): Recommended Phase 2 Dose (RP2D) of Orally Administered THE-630
Description: The RP2D was expected to be equal to the MTD or less than the MTD, if aspects of tolerability or efficacy not encompassed by the MTD determination suggested utilizing a lower dose.
Time Frame: 28 days
Population: as for outcome 2
Measure: Number; unit: mg
Arm/Group | Dose Escalation (3 mg to 27 mg Once Daily)
Number analyzed (Participants) | 27
mg | NA — The RP2D was not determined, in part because the MTD could not be identified. The study was terminated by the Sponsor due to dose-limiting toxicities prior to initiation of the Expansion phase (Phase 2) of the study.

5. Primary Outcome: Expansion (Phase 2): Efficacy Assessment - For Each Expansion Phase Cohort (Cohorts 1, 2, and 3), Confirmed Objective Response Rate (ORR), According to Modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1
Time Frame: Up to 24 months after first dose
Population: The Sponsor terminated the study due to early dose-limiting toxicities and not initiate Expansion Cohort 1, Expansion Cohort 2 or Expansion Cohort 3 (Phase 2).
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Dose Escalation (Phase 1): Plasma Pharmacokinetic (PK) Parameters of THE-630 and Its Active Metabolite - Cmax (Maximum Observed Concentration)
Description: Cmax of THE-630 and its active metabolite after single oral dose and at steady state after multiple oral doses
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 28 days)
Population: The scope of planned analyses and data reporting was reduced (per statistical analysis plan [SAP] v3.0), given the Sponsor's decision to terminate the study early due to dose-limiting toxicities and to discontinue the THE-630 development program. As a result, data for this outcome measure are not available.
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Dose Escalation (Phase 1): Plasma PK Parameters of THE-630 and Its Active Metabolite - Tmax (Time of First Occurrence of Cmax)
Description: Tmax of THE-630 and its active metabolite after single oral dose and at steady state after multiple oral doses
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 28 days)
Population: The scope of planned analyses and data reporting was reduced (per SAP v3.0), given the Sponsor's decision to terminate the study early due to dose-limiting toxicities and to discontinue the THE-630 development program. As a result, data for this outcome measure are not available.
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Dose Escalation (Phase 1): Plasma PK Parameters of THE-630 and Its Active Metabolite - AUC 0-24 (Area Under the Concentration-time Curve From Time Zero to 24 Hours)
Description: AUC 0-24 of THE-630 and its active metabolite after single oral dose and at steady state after multiple oral doses
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 28 days)
Population: as for outcome 7
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Dose Escalation (Phase 1): Plasma PK Parameters of THE-630 and Its Active Metabolite - AUC 0-t (Area Under the Concentration-time Curve From Time Zero to Time t)
Description: AUC 0-t of THE-630 and its active metabolite after single oral dose and at steady state after multiple oral doses
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 28 days)
Population: as for outcome 7
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Dose Escalation (Phase 1): Efficacy Assessment - Confirmed ORR, According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: Full Analysis Set, which includes all patients who were enrolled and received at least 1 dose of THE-630.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 7 | 6
percentage of participants | 0 [0 to 70.8] | 0 [0 to 41.0] | 0 [0 to 70.8] | 0 [0 to 70.8] | 0 [0 to 70.8] | 0 [0 to 41.0] | 0 [0 to 45.9]

11. Secondary Outcome: Dose Escalation (Phase 1): Efficacy Assessment - Best Overall Response, According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: Full Analysis Set, which includes all patients who were enrolled and received at least 1 dose of THE-630.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 7 | 6
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Parital Response (PR) | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Stable Disease (SD) | 0 | 1 | 1 | 3 | 3 | 3 | 4
  Progressive Disease (PD) | 3 | 3 | 2 | 0 | 0 | 3 | 2
  Not Evaluable (NE) | 0 | 3 | 0 | 0 | 0 | 1 | 0

12. Secondary Outcome: Dose Escalation (Phase 1): Efficacy Assessment - Best Target Lesion Response, According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: as for outcome 7
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Dose Escalation (Phase 1): Efficacy Assessment - Time to Response, According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: as for outcome 7
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Dose Escalation (Phase 1): Efficacy Assessment - Duration of Response (DOR), According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: as for outcome 7
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Dose Escalation (Phase 1): Efficacy Assessment - Disease Control Rate (DCR), According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: Full Analysis Set, which includes all patients who were enrolled and received at least 1 dose of THE-630.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 7 | 6
percentage of participants | 0 [0 to 70.8] | 14.3 [0.4 to 57.9] | 33.3 [0.8 to 90.6] | 100 [29.2 to 100] | 100 [29.2 to 100] | 42.9 [9.9 to 81.6] | 66.7 [22.3 to 95.7]

16. Secondary Outcome: Dose Escalation (Phase 1): Efficacy Assessment - Clinical Benefit Rate (CBR) at 16 Weeks, According to Modified RECIST 1.1
Time Frame: 16 weeks
Population: Full Analysis Set, which includes all patients who were enrolled and received at least 1 dose of THE-630.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3 | 7 | 6
percentage of participants | 0 [0 to 70.8] | 14.3 [0.4 to 57.9] | 0 [0 to 70.8] | 66.7 [9.4 to 99.2] | 66.7 [9.4 to 99.2] | 14.3 [0.4 to 57.9] | 50.0 [11.8 to 88.2]

17. Secondary Outcome: Dose Escalation (Phase 1): Efficacy Assessment - Progression Free Survival (PFS), According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: as for outcome 7
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Dose Escalation (Phase 1): Efficacy Assessment - Overall Survival (OS)
Time Frame: Up to 24 months after first dose
Population: as for outcome 7
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Expansion (Phase 2): Efficacy Assessment - Best Overall Response, According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

20. Secondary Outcome: Expansion (Phase 2): Efficacy Assessment - Best Target Lesion Response, According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

21. Secondary Outcome: Expansion (Phase 2): Efficacy Assessment - Time to Response, According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

22. Secondary Outcome: Expansion (Phase 2): Efficacy Assessment - DOR, According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

23. Secondary Outcome: Expansion (Phase 2): Efficacy Assessment - DCR, According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

24. Secondary Outcome: Expansion (Phase 2): Efficacy Assessment - CBR at 16 Weeks, According to Modified RECIST 1.1
Time Frame: 16 weeks
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

25. Secondary Outcome: Expansion (Phase 2): Efficacy Assessment - PFS, According to Modified RECIST 1.1
Time Frame: Up to 24 months after first dose
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

26. Secondary Outcome: Expansion (Phase 2): Efficacy Assessment - OS
Time Frame: Up to 24 months after first dose
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

27. Secondary Outcome: Expansion (Phase 2): Safety Analysis - Number of Participants With Treatment-emergent Adverse Events as Assessed by NCI CTCAE v5.0
Time Frame: Up to 24 months after first dose
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

28. Secondary Outcome: Expansion (Phase 2): Plasma PK Parameters of THE-630 and Its Active Metabolite - Cmax (Maximum Observed Concentration)
Description: Cmax of THE-630 and its active metabolite after single oral dose and at steady state after multiple oral doses
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 28 days)
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

29. Secondary Outcome: Expansion (Phase 2): Plasma PK Parameters of THE-630 and Its Active Metabolite - Tmax (Time of First Occurrence of Cmax)
Description: Tmax of THE-630 and its active metabolite after single oral dose and at steady state after multiple oral doses
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 28 days)
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

30. Secondary Outcome: Expansion (Phase 2): Plasma PK Parameters of THE-630 and Its Active Metabolite - AUC 0-24 (Area Under the Concentration-time Curve From Time Zero to 24 Hours)
Description: AUC 0-24 of THE-630 and its active metabolite after single oral dose and at steady state after multiple oral doses
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 28 days)
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

31. Secondary Outcome: Expansion (Phase 2): Plasma PK Parameters of THE-630 and Its Active Metabolite - AUC 0-t (Area Under the Concentration-time Curve From Time Zero to Time t)
Description: AUC 0-t of THE-630 and its active metabolite after single oral dose and at steady state after multiple oral doses
Time Frame: Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 28 days)
Population: as for baseline characteristics
Arm/Group | Expansion Cohort 1 | Expansion Cohort 2 | Expansion Cohort 3
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 24 months after first dose
Description: Dose Escalation (Phase 1): Safety Analysis - Number of participants with treatment-emergent adverse events as assessed by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Arm/Group | Dose Escalation (3 mg Once Daily) | Dose Escalation (4 mg Once Daily) | Dose Escalation (6 mg Once Daily) | Dose Escalation (9 mg Once Daily) | Dose Escalation (12 mg Once Daily) | Dose Escalation (18 mg Once Daily) | Dose Escalation (27 mg Once Daily)
All-Cause Mortality (participants affected / at risk) | 3/3 | 6/7 | 2/3 | 0/3 | 1/3 | 2/7 | 1/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 5/7 | 1/3 | 0/3 | 1/3 | 5/7 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 3/3 | 3/3 | 3/3 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation (3 mg Once Daily) (N=3) | Dose Escalation (4 mg Once Daily) (N=7) | Dose Escalation (6 mg Once Daily) (N=3) | Dose Escalation (9 mg Once Daily) (N=3) | Dose Escalation (12 mg Once Daily) (N=3) | Dose Escalation (18 mg Once Daily) (N=7) | Dose Escalation (27 mg Once Daily) (N=6)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Escalation (3 mg Once Daily) (N=3) | Dose Escalation (4 mg Once Daily) (N=7) | Dose Escalation (6 mg Once Daily) (N=3) | Dose Escalation (9 mg Once Daily) (N=3) | Dose Escalation (12 mg Once Daily) (N=3) | Dose Escalation (18 mg Once Daily) (N=7) | Dose Escalation (27 mg Once Daily) (N=6)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 1 | 0 | 1 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 2 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 2 | 4
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2 | 2 | 2
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Saliva altered (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 2 | 1 | 2 | 2 | 3
Oedema peripheral (General disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0
Thirst (General disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Early satiety (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 0 | 0 | 1 | 0 | 4 | 2
Weight decreased (Investigations) | 1 | 1 | 1 | 0 | 1 | 1 | 2
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 3 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 2 | 2
Amylase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 4
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 1 | 1 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Trigeminal nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Libido decreased (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oedema genital (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 3 | 0 | 0 | 0 | 1 | 4 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
The Sponsor made a business decision to terminate the trial early due to observed dose limiting toxicities at dose levels that are below the target THE-630 exposure (set by preclinical studies) required for pan KIT variant inhibition in GIST patients. Therefore, several of the outcome measures could not be evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements between Theseus Pharmaceuticals and individual investigators may vary. Theseus has the right to review results disclosures prior to public release and can embargo results disclosures for >60 days but ≤180 days from the date of submission for review. Theseus supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-12-07): https://cdn.clinicaltrials.gov/large-docs/68/NCT05160168/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/68/NCT05160168/SAP_001.pdf